CLINICAL TRIAL: NCT05443841
Title: A Prospective Study for Pleural Lavage Cytology in Patients With Esophageal Cancer
Brief Title: Value of Pleural Lavage Cytology in Resectable Esophageal Carcinoma Eastern Cooperative Thoracic Oncology Projects 2005, ECTOP-2005)
Acronym: ECTOP-2005
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Fudan University Shanghai Cancer Center, Fudan University
Other Study IDs: ECTOP-2005
Record Dates: First submitted 2022-06-22; First posted 2022-07-05 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Esophageal Cancer
Keywords: Squamous cell carcinoma; Esophagectomy; Pleural Lavage
MeSH Terms: conditions — Esophageal Neoplasms; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: pleural lavage — pleural lavages before tumor resection and after tumor resecion, respectively

SUMMARY:
Disease recurrence and metastasis are common after curative treatment for patients with esophageal cancer. Thus, it is important to identify the risk factors to predict disease recurrence and metastasis. Pleural lavage cytology (PLC) is reported to be associated with disease recurrence and patient survival in lung cancer, but the value is unclear in esophageal cancer. The aim of this study is to evaluate the value of PLC in esophageal cancer patient in terms of frequencies, association with patient survival, and efficacy of postoperative treatment.

DETAILED DESCRIPTION:
Pleural lavage cytology will be performed before esophageal resection, and after resection, respectively. Frequency of positive pleural lavage cytology will be determined, and the value of pleural lavage cytology for patients with resectable esophageal cancer will be studied.

ELIGIBILITY:
Inclusion Criteria:

* esophageal cancer with histological confirmation before treatment.
* resectable esophageal cancer with clinical T1-4a/N0-3/M0 staging
* potential R0 resection
* no history of other malignancies

Exclusion Criteria:

* severe major organ dysfunction (American society of anesthesiologisits score >3 )
* patients underwent ESD or EMR
* pleural lavage is unavailable due to adhesions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with esophageal cancer
Sampling Method: Probability Sample
Enrollment: 385 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
number of patients who had positive pleural lavage cytology | July 2022 to July 2023
  Frequency of positive pleural lavage cytology in resectable esophageal squamous cell carcinoma

SECONDARY OUTCOMES:
Time period from date of surgery to the date of death | July 2022 to July 2026
  value of pleural lavage cytology in predict patient survival

CONTACTS AND LOCATIONS:
Overall Officials: Haiquan Chen, MD, Principal Investigator — Fudan University
Locations (11):
- China (11):
  - The First Affiliated Hospital of USTC, Hefei, Anhui
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - The Second Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Taixing People's Hospital, Taishing, Jiangsu
  - Taizhou People's Hospital, Taizhou, Jiangsu
  - Shaanxi Provincial cancer Hospital, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shannxi
  - Tianjin Medical University Cancer Institute, Tianjin, Tianjin Municipality
  - Fudan University Shanghai Cancer Center, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided
individual participant data could be shared after the recruitment of all 385 patients